CLINICAL TRIAL: NCT05282771
Title: A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study, Comparing Halobetasol Propionate and Tazarotene Topical Lotion 0.01%/0.045% (Taro Pharmaceuticals U.S.A., Inc.) to Duobrii® Lotion (Halobetasol Propionate and Tazarotene Lotion), 0.01%/0.045% (Reference Listed Drug) and Both Active Treatments to a Placebo Control in the Treatment of Moderate to Severe Plaque Psoriasis
Brief Title: A Study Comparing Halobetasol Propionate and Tazarotene Topical Lotion 0.01%/0.045% to Duobrii® Lotion (Halobetasol Propionate and Tazarotene Lotion), 0.01%/0.045% (Reference Listed Drug) in the Treatment of Moderate to Severe Plaque Psoriasis.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLBT-2001
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — halobetasol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Halobetasol Propionate and Tazarotene Topical lotion 0.01%/0.045% (Experimental): The study drug is to be self-administered by applying as a thin layer once daily to cover only affected areas and rubbed in gently for approximately 8 weeks
  Interventions: Drug: Halobetasol Propionate and Tazarotene Lotion 0.01%/0.045%
- Duobrii® Lotion (Halobetasol propionate and tazarotene lotion), 0.01%/0.045% (Active Comparator): The study drug is to be self-administered by applying as a thin layer once daily to cover only affected areas and rubbed in gently for approximately 8 weeks
  Interventions: Drug: Duobrii® Lotion (Halobetasol propionate and tazarotene lotion), 0.01%/0.045%
- Placebo Control (Placebo Comparator): The study drug is to be self-administered by applying as a thin layer once daily to cover only affected areas and rubbed in gently for approximately 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Halobetasol Propionate and Tazarotene Lotion 0.01%/0.045% — The study drug is to be self-administered by applying as a thin layer once daily to cover only affected areas and rubbed in gently for approximately 8 weeks.
  Other Names: Test Product
  Arms: Halobetasol Propionate and Tazarotene Topical lotion 0.01%/0.045%
Drug: Duobrii® Lotion (Halobetasol propionate and tazarotene lotion), 0.01%/0.045% — The study drug is to be self-administered by applying as a thin layer once daily to cover only affected areas and rubbed in gently for approximately 8 weeks.
  Other Names: Reference Product
  Arms: Duobrii® Lotion (Halobetasol propionate and tazarotene lotion), 0.01%/0.045%
Drug: Placebo — The study drug is to be self-administered by applying as a thin layer once daily to cover only affected areas and rubbed in gently for approximately 8 weeks.
  Other Names: Vehicle
  Arms: Placebo Control

SUMMARY:
To evaluate the therapeutic equivalence and safety of halobetasol propionate and tazarotene topical lotion 0.01%/0.045% (Taro Pharmaceuticals U.S.A., Inc.) and Duobrii® Lotion (halobetasol and tazarotene lotion), 0.01%/0.045% (Reference Listed Drug) in the treatment of moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
A Multi-center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study, Comparing Halobetasol Propionate and Tazarotene Topical Lotion 0.01%/0.045% (Taro Pharmaceuticals U.S.A., Inc.) and Duobrii® Lotion (Halobetasol propionate and tazarotene lotion), 0.01%/0.045% (Reference Listed Drug) in the Treatment of Moderate to Severe Plaque Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 18 years
* Subjects must have provided IRB approved written informed consent
* Subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits
* Subjects with a clinical diagnosis of stable (at least 6 months) plaque psoriasis involving at least 3% and no more than 12% of the body surface area (BSA). Affected areas should not include the axillae, face, scalp, soles, palms, and intertriginous areas

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Females of childbearing potential who do not agree to utilize an adequate form of contraception.
* Subjects with a known hypersensitivity to tazarotene, halobetasol propionate, other corticosteroids, or to any ingredients in the study drugs.
* Subjects with current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects with a response of "treatment success" on the IGA of disease severity at Week 8 | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Zaidoon A. Al-Zubaidy, Study Director — Catawba Research
Locations (1):
- Catawba Research, LLC, Charlotte, North Carolina, United States